

Date

## **Consent Form**

\_\_\_\_\_

## Title of Project

The role of cardiopulmonary exercise testing in the diagnosis and management of people with Heart Failure.

| <b>Name of Principal Investigator:</b> Dr. Peter McKavanagh | | | |
|---|---|---|---|
| Please initial | | | |
| • I confirm that I have read and understood the have had the opportunity to consider the informatisfactorily. | - | | - |
| | | [Initial here: | ] |
| • I understand that my participation is voluntary, a reason and without any effect on the healthca | | | ing |
| <ul> <li>I understand that relevant sections of my medilooked at by researchers from Ulster University taking part in this research. I give permission for</li> <li>I understand that the information held and medical contents.</li> </ul> | and from the NHS Trust, where these individuals to have access | e it is relevant to it to my records. [Initial here: | my<br>] |
| used to help contact me or provide information | • | iai care trust may | שפ |
| | | [Initial here: | ] |
| • I agree to take part in the above study. | | [Initial here: | ] |
| Name participant | Signature | Date | |
| | | | _ |

Please return one signed copy of this form to the Chief Investigator. Please retain the other copy for your records. If you have any questions about the study or should you require any additional information please contact:

Signature

Dr. Peter McKavanagh Cardiology Dept, Ulster Hospital, Dundonald Secretary Tel: 028 9048 4511 ext 21762 Email: Wendy.Wratten@setrust.hscni.net

Name of researcher

One copy for the participant; one copy for the researcher.